CLINICAL TRIAL: NCT06473935
Title: Maternal Well-being in the Perinatal Period: a Prospective Observational Study
Brief Title: Maternal Well-being in the Perinatal Period
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Valentina Di Mattei, Professor, IRCCS San Raffaele
Other Study IDs: Benessere Materno23
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Perinatal Depression; Anxiety; Loneliness; Mother-Child Relations
MeSH Terms: conditions — Anxiety Disorders | interventions — Surveys and Questionnaires; Focus Groups

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women during pregnancy and postpartum: Women during the last trimester of gestation (28th-35th week of gestation) and during the 18 months following the child's birth
  Interventions: Other: Questionnaires and focus groups

INTERVENTIONS:
Other: Questionnaires and focus groups — Participation in the research involves completing a test battery composed of self-administered questionnaires, all validated in the Italian language.
  Additionally, qualitative data will be collected through semi-structured interviews (conducted in person or online, based on individual preferences) and focus groups, both lasting between 90 and 120 minutes.

SUMMARY:
The goal of this observation study is to investigate the mental health status of women experiencing their first pregnancy, with particular attention to anxiety and depression symptoms, feelings of loneliness, and the quality of defense mechanisms employed.

DETAILED DESCRIPTION:
The primary goal of this observational study si to investigate the mental health status of women experiencing their first pregnancy, with particular attention to manifestations of anxiety and depression, feelings of loneliness, and the quality of defense mechanisms employed, during the last trimester of gestation (28th-35th week of gestation) and over the course of the 18 months following the child's birth.

Furthermore, the study aims to conduct an in-depth analysis of the variables associated with the psychological adaptation of women during the perinatal period, with particular reference to the following exploratory objectives:

* To explore the association between the investigated psychological dimensions and the quality of the bond with the child in the prenatal and postnatal periods.
* To identify any significant differences in the variables of interest between women who conceived naturally and those who underwent assisted reproductive technology (ART).
* To detect, through qualitative methods (semi-structured interviews and focus groups), the unmet needs of women during the perinatal period, as well as their preferences and expectations regarding the nature of desirable support interventions during this period. This would enable the construction and provision of an intervention model that closely aligns with the specific needs of this patient population.

The collected data will allow for the identification of individuals at higher risk of psychological distress and adaptation problems during the perinatal period, as well as potential impairment in the quality of the attachment bond with the child.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Adequate understanding of the Italian language
* Willingness to participate in the study, expressed through the signing of the information sheet, consent declaration, and privacy statement
* Women experiencing their first pregnancy
* Women in the last trimester of gestation (28th-35th week of gestation) who will be followed for 18 months after childbirth

Exclusion Criteria:

* Age under 18 years old
* Women who are not able to understand the Italian language
* Absence of the willingness to participate in the study, expressed through the signing of the information sheet, consent declaration, and privacy statement
* Women who are not experiencing their first pregnancy
* Women who are not in the last trimester of gestation (28th-35th week of gestation)

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: We plan to recruit a sample of at least 134 patients. This sample size allows us to meet the recommendations obtained from conducting the power analysis.
  The sample size calculation was performed using G*Power software (version 3.1.9.6, Faul et al., 2007).
Sampling Method: Non-Probability Sample
Enrollment: 134 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Depression | June 1, 2024 - December 31, 2025
  Levels of perinatal depression and of pregnancy-related anxiety
Anxiety | June 1, 2024 - December 31, 2025
  Levels of state and trait anxiety
Loneliness | June 1, 2024 - December 31, 2025
  Feelings of loneliness during and after pregnancy
Defense mechanisms | June 1, 2024 - December 31, 2025
  Nature of defense mechanisms during and after pregnancy

SECONDARY OUTCOMES:
Attachment bond | June 1, 2024 - December 31, 2025
  Quality of prenatal of attachment bond and in the postpartum period
Women subjective experience | June 1, 2024 - December 31, 2025
  Subjective experience of pregnancy and postpartum
Unmet needs of women | June 1, 2024 - December 31, 2025
  Unmet needs of women during the perinatal period

CONTACTS AND LOCATIONS:
Overall Officials: Valentina Di Mattei, Professor, Principal Investigator — IRCCS San Raffaele
Locations (1):
- IRCCS San Raffaele, Milan, Italy